CLINICAL TRIAL: NCT01198756
Title: Immunogenicity and Safety Study of GSK Biologicals' Quadrivalent Influenza Vaccine (GSK2282512A) When Administered in Children
Brief Title: A Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Seasonal Influenza Vaccine in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 113314
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-04

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- GSK2282512A 1 Group (Experimental): Subjects, 3 to 17 years old, received 1 dose of GSK2282512A vaccine at Day 0 or 2 doses of GSK2282512A vaccine at Day 0 and Day 28. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Quadrivalent seasonal influenza vaccine GSK2282512A
- Victoria strain Fluarix Group (Active Comparator): Subjects, 3 to 17 years old, received 1 dose of Fluarix™ VB vaccine containing the Victoria lineage B flu strain at Day 0 or 2 doses of Fluarix™ VB vaccine at Day 0 and Day 28. The Fluarix™ VB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix™ VB
- Yamagata strain Fluarix Group (Active Comparator): Subjects, 3 to 17 years old, received 1 dose of Fluarix™ YB vaccine containing the Yamagata lineage B flu strain at Day 0 or 2 doses of Fluarix™ YB vaccine at Day 0 and Day 28. The Fluarix™ YB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix™ YB
- GSK2282512A 2 Group (Experimental): Subjects, 6 to 35 months old, received 1 dose of GSK2282512A vaccine at Day 0 or 2 doses of GSK2282512A vaccine at Day 0 and Day 28. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm for subjects ≥12 months of age and into the antero-lateral region of the left thigh for infants <12 months of age.
  Interventions: Biological: Quadrivalent seasonal influenza vaccine GSK2282512A

INTERVENTIONS:
Biological: Quadrivalent seasonal influenza vaccine GSK2282512A — For subject 3 to 8 years of age, single intramuscular dose for primed subjects, two doses for unprimed subjects. For subjects 9 to 17 years of age, single intramuscular dose.
  Arms: GSK2282512A 1 Group
Biological: Fluarix™ VB — For subject 3 to 8 years of age, single intramuscular dose for primed subjects, two doses for unprimed subjects. For subjects of 9 to 17 years of age, single intramuscular dose.
  Arms: Victoria strain Fluarix Group
Biological: Fluarix™ YB — For subject 3 to 8 years of age, single intramuscular dose for primed subjects, two doses for unprimed subjects. For subjects of 9 to 17 years of age, single intramuscular dose
  Arms: Yamagata strain Fluarix Group
Biological: Quadrivalent seasonal influenza vaccine GSK2282512A — Single intramuscular dose for primed subjects, two doses for unprimed subjects.
  Arms: GSK2282512A 2 Group

SUMMARY:
This study is designed to test the immunogenicity and safety of an investigational influenza vaccine, in children compared to two other influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parent(s) or legally acceptable representative(s) can and will comply with the requirements of the protocol.
* A male or female child aged between 6 months and 17 years inclusive at the time of the first vaccination; children are eligible regardless of history of administration of influenza vaccine in a previous season.
* Written informed consent obtained from the subject/from the parent(s)/legally acceptable representative(s) of the subject.
* Written informed assent obtained from the subject if/as required by local regulations.
* Subjects in stable health as determined by investigator's clinical examination and assessment of subjects' medical history.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject

  * Has practiced adequate contraception for 30 days prior to vaccination, and
  * Has a negative pregnancy urine test on the day of vaccination, and
  * Has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Child in care
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.Prior receipt of any seasonal or pandemic influenza vaccine within 6 months preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune modifying drugs within six months prior to the first vaccine dose.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* History of Guillain-Barré syndrome within 6 weeks of receipt of prior influenza vaccine.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Fever at the time of enrolment.
* Acute disease at the time of enrolment.
* Any significant disorder of coagulation or treatment with Coumadin derivatives or heparin.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Ongoing aspirin therapy.
* Any other condition which, in the opinion of the Investigator, prevents the subject from participating in the study.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3109 (Actual)
Dates: Start 2010-10-01; Primary Completion 2011-07-01 (Actual); Study Completion 2011-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- United States (16):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Harrisburg, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Thornton, Colorado
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Barnwell, South Carolina
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Fort Worth, Texas
- Canada (9):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Mount Pearl, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Saskatoon, Saskatchewan
- Mexico (2):
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Mexico City
- Spain (4):
  - GSK Investigational Site, Alcalá de Guadaira
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Seville
- Taiwan (2):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Langley JM, Carmona Martinez A, Chatterjee A, Halperin SA, McNeil S, Reisinger KS, Aggarwal N, Huang LM, Peng CT, Garcia-Sicilia J, Salamanca de la Cueva I, Cabanas F, Trevino-Garza C, Rodriguez-Weber MA, de la O M, Chandrasekaran V, Dewe W, Liu A, Innis BL, Jain VK. Immunogenicity and safety of an inactivated quadrivalent influenza vaccine candidate: a phase III randomized controlled trial in children. J Infect Dis. 2013 Aug 15;208(4):544-53. doi: 10.1093/infdis/jit263. Epub 2013 Jul 11. PMID 23847058
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 113314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 3109 subjects were enrolled, out of which solely 3094 subjects were vaccinated who constituted the analysed population in this study.
Pre-assignment Details: Unprimed Subjects - subjects aged 6 months to 8 years with no H1N1 vaccine or H1N1 infection in the last season, or with no seasonal influenza vaccine in the past or who had received only 1 dose for the first time in the last season - received a 2-dose vaccination course. Primed Subjects - all other subjects - received a 1-dose vaccination course.
Period: Overall Study
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Started | 932 | 929 | 932 | 301
Completed | 894 | 889 | 902 | 275
Not Completed | 38 | 40 | 30 | 26
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 9 | 4 | 7 | 5
Not completed — Lost to Follow-up | 29 | 36 | 23 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group | Total
Number analyzed (Participants) | 932 | 929 | 932 | 301 | 3094
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.9 (4.21) | 8.9 (4.23) | 8.9 (4.17) | 1.2 (0.73) | 8.1 (4.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 434 | 455 | 464 | 143 | 1496
  Male | 498 | 474 | 468 | 158 | 1598

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was the seropositivity cut-off of 1:10. Antibodies assessed were antibodies against the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Florida/4/2006 (Yamagata) flu strains.
Time Frame: At 28 days after administration of the last vaccine dose (Day 28 for Primed Subjects and at Day 56 for Unprimed Subjects) (POST)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable and eligible subjects for whom data concerning immunogenicity outcomes variables were available and for whom assay results were available for antibodies against at least one study vaccine component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 878 | 871 | 878 | 259
titer
  H1N1, POST | 362.7 [335.3 to 392.3] | 429.1 [396.5 to 464.3] | 420.2 [388.8 to 454.0] | 200.9 [166.6 to 242.2]
  H3N2, POST | 143.7 [134.2 to 153.9] | 139.6 [130.5 to 149.3] | 151.0 [141.0 to 161.6] | 61.4 [53.8 to 70.0]
  Victoria, POST: number analyzed (Participants) | 878 | 871 | 877 | 259
  Victoria, POST | 250.5 [230.8 to 272.0] | 245.4 [226.9 to 265.4] | 68.1 [61.9 to 74.9] | 127.3 [109.4 to 148.1]
  Yamagata, POST | 512.5 [477.6 to 549.9] | 197.0 [180.7 to 214.8] | 579.0 [541.2 to 619.3] | 192.7 [172.1 to 215.7]

2. Primary Outcome: Number of Subjects Seroconverted Against 4 Strains of Influenza Disease
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥1:40, or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The vaccine strains assessed were the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Florida/4/2006 (Yamagata) flu strains.
Time Frame: as for outcome 1
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, inclusive of all evaluable and eligible subjects with immunogenicity results available for antibodies against at least one study vaccine component after vaccination, solely on subjects with both pre- and post-vaccination immunogenicity results available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 876 | 870 | 877 | 259
Participants
  H1N1, POST | 739 | 755 | 750 | 220
  H3N2, POST: number analyzed (Participants) | 876 | 870 | 876 | 259
  H3N2, POST | 614 | 590 | 610 | 189
  Victoria, POST: number analyzed (Participants) | 876 | 870 | 876 | 259
  Victoria, POST | 653 | 622 | 262 | 219
  Yamagata, POST | 659 | 359 | 644 | 243

3. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease
Description: as for outcome 1
Time Frame: At Day 0 and at 28 days after administration of the last vaccine dose (Day 28 for Primed Subjects and at Day 56 for Unprimed Subjects) (POST)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 878 | 871 | 878 | 259
titer
  H1N1, Day 0: number analyzed (Participants) | 876 | 870 | 877 | 259
  H1N1, Day 0 | 29.4 [26.8 to 32.2] | 32.2 [29.4 to 35.3] | 29.1 [26.6 to 31.8] | 16.8 [13.9 to 20.3]
  H1N1, POST | 362.7 [335.3 to 392.3] | 429.1 [396.5 to 464.3] | 420.2 [388.8 to 454.0] | 200.9 [166.6 to 242.2]
  H3N2, Day 0: number analyzed (Participants) | 876 | 870 | 876 | 259
  H3N2, Day 0 | 18.1 [16.7 to 19.7] | 19.0 [17.4 to 20.6] | 19.4 [17.8 to 21.1] | 5.6 [5.3 to 6.0]
  H3N2, POST | 143.7 [134.2 to 153.9] | 139.6 [130.5 to 149.3] | 151.0 [141.0 to 161.6] | 61.4 [53.8 to 70.0]
  Victoria, Day 0: number analyzed (Participants) | 876 | 870 | 877 | 259
  Victoria, Day 0 | 24.8 [22.5 to 27.3] | 25.8 [23.5 to 28.4] | 25.8 [23.5 to 28.4] | 8.7 [7.5 to 10.0]
  Victoria, POST: number analyzed (Participants) | 878 | 871 | 877 | 259
  Victoria, POST | 250.5 [230.8 to 272.0] | 245.4 [226.9 to 265.4] | 68.1 [61.9 to 74.9] | 127.3 [109.4 to 148.1]
  Yamagata, Day 0: number analyzed (Participants) | 876 | 870 | 877 | 259
  Yamagata, Day 0 | 57.9 [52.0 to 64.4] | 58.4 [52.6 to 64.9] | 65.9 [59.3 to 73.2] | 7.7 [7.0 to 8.6]
  Yamagata, POST | 512.5 [477.6 to 549.9] | 197.0 [180.7 to 214.8] | 579.0 [541.2 to 619.3] | 192.7 [172.1 to 215.7]

4. Secondary Outcome: Number of Subjects Seroprotected Against 4 Strains of Influenza Disease
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition titer ≥ 1:40. The 4 assessed influenza strains were the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Florida/4/2006 flu strains.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 878 | 871 | 878 | 259
Participants
  H1N1, Day 0: number analyzed (Participants) | 876 | 870 | 877 | 259
  H1N1, Day 0 | 480 | 496 | 477 | 87
  H1N1, POST | 850 | 848 | 848 | 232
  H3N2, Day 0: number analyzed (Participants) | 876 | 870 | 876 | 259
  H3N2, Day 0 | 295 | 301 | 324 | 7
  H3N2, POST | 816 | 808 | 819 | 193
  Victoria, Day 0: number analyzed (Participants) | 876 | 870 | 877 | 259
  Victoria, Day 0 | 388 | 404 | 400 | 28
  Victoria, POST: number analyzed (Participants) | 878 | 871 | 877 | 259
  Victoria, POST | 838 | 839 | 643 | 228
  Yamagata, Day 0: number analyzed (Participants) | 876 | 870 | 877 | 259
  Yamagata, Day 0 | 578 | 583 | 622 | 22
  Yamagata, POST | 869 | 805 | 873 | 250

5. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination (at Day 28 for Primed Subjects and at Day 56 for Unprimed Subjects (POST)) compared to Day 0 (i.e. the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer). The 4 assessed influenza strains were the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Florida/4/2006 (Yamagata) flu strains
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 876 | 870 | 877 | 259
fold change
  H1N1, POST | 12.31 [11.34 to 13.35] | 13.31 [12.28 to 14.43] | 14.42 [13.27 to 15.66] | 11.95 [10.52 to 13.59]
  H3N2, POST: number analyzed (Participants) | 876 | 870 | 876 | 259
  H3N2, POST | 7.94 [7.30 to 8.64] | 7.37 [6.78 to 8.02] | 7.78 [7.16 to 8.46] | 10.94 [9.64 to 12.42]
  Victoria, POST: number analyzed (Participants) | 876 | 870 | 876 | 259
  Victoria, POST | 10.12 [9.23 to 11.09] | 9.51 [8.64 to 10.45] | 2.63 [2.47 to 2.81] | 14.61 [12.84 to 16.63]
  Yamagata, POST | 8.86 [8.12 to 9.66] | 3.37 [3.14 to 3.62] | 8.78 [8.05 to 9.58] | 24.92 [21.98 to 28.26]

6. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease - By Age Strata
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was the seropositivity cut-off of 1:10. Antibodies assessed were antibodies against the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Florida/4/2006 (Yamagata) flu strains. Subjects were assessed according to 3 age categories, 3-8 years, 9-17 years and 6-35 months.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- GSK2282512A 1 (3-8 Years) Group: Subjects, 3 to 8 years old, received 1 dose of GSK2282512A vaccine at Day 0 or 2 doses of GSK2282512A vaccine at Day 0 and Day 28. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- GSK2282512A 1 (9-17 Years) Group: Subjects, 9 to 17 years old, received 1 dose of GSK2282512A vaccine at Day 0 or 2 doses of GSK2282512A vaccine at Day 0 and Day 28. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Victoria Strain Fluarix (3-8 Years) Group: Subjects, 3 to 8 years old, received 1 dose of Fluarix™ VB vaccine containing the Victoria lineage B flu strain at Day 0 or 2 doses of Fluarix™ VB vaccine at Day 0 and Day 28. The Fluarix™ VB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Victoria Strain Fluarix (9-17 Years) Group: Subjects, 9 to 17 years old, received 1 dose of Fluarix™ VB vaccine containing the Victoria lineage B flu strain at Day 0 or 2 doses of Fluarix™ VB vaccine at Day 0 and Day 28. The Fluarix™ VB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Yamagata Strain Fluarix (3-8 Years) Group: Subjects, 3 to 8 years old, received 1 dose of Fluarix™ YB vaccine containing the Yamagata lineage B flu strain at Day 0 or 2 doses of Fluarix™ YB vaccine at Day 0 and Day 28. The Fluarix™ YB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Yamagata Strain Fluarix (9-17 Years) Group: Subjects, 9 to 17 years old, received 1 dose of Fluarix™ YB vaccine containing the Yamagata lineage B flu strain at Day 0 or 2 doses of Fluarix™ YB vaccine at Day 0 and Day 28. The Fluarix™ YB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | GSK2282512A 1 (3-8 Years) Group | GSK2282512A 1 (9-17 Years) Group | Victoria Strain Fluarix (3-8 Years) Group | Victoria Strain Fluarix (9-17 Years) Group | Yamagata Strain Fluarix (3-8 Years) Group | Yamagata Strain Fluarix (9-17 Years) Group | GSK2282512A 2 Group
Number analyzed (Participants) | 425 | 453 | 424 | 447 | 424 | 454 | 259
titer
  H1N1, Day 0: number analyzed (Participants) | 423 | 453 | 423 | 447 | 424 | 453 | 259
  H1N1, Day 0 | 24.7 [21.6 to 28.3] | 34.6 [30.6 to 39.2] | 26.9 [23.5 to 30.9] | 38.2 [33.8 to 43.1] | 24.5 [21.5 to 27.8] | 34.2 [30.3 to 38.6] | 16.8 [13.9 to 20.3]
  H1N1, POST | 310.5 [274.9 to 350.6] | 419.5 [379.8 to 463.4] | 382.7 [339.4 to 431.6] | 478.2 [431.4 to 530.0] | 356.2 [316.5 to 400.8] | 490.3 [443.7 to 541.7] | 200.9 [166.6 to 242.2]
  H3N2, Day 0: number analyzed (Participants) | 423 | 453 | 423 | 447 | 423 | 453 | 259
  H3N2, Day 0 | 19.7 [17.4 to 22.4] | 16.7 [15.0 to 18.7] | 21.2 [18.6 to 24.2] | 17.0 [15.3 to 19.0] | 20.2 [17.8 to 23.0] | 18.6 [16.6 to 20.9] | 5.6 [5.3 to 6.0]
  H3N2, POST | 138.2 [123.7 to 154.5] | 149.1 [137.3 to 162.0] | 144.4 [130.6 to 159.7] | 135.2 [123.5 to 148.0] | 147.9 [133.3 to 164.1] | 153.9 [140.7 to 168.4] | 61.4 [53.8 to 70.0]
  Victoria, Day 0: number analyzed (Participants) | 423 | 453 | 423 | 447 | 424 | 453 | 259
  Victoria, Day 0 | 18.3 [15.8 to 21.1] | 32.9 [29.0 to 37.4] | 20.2 [17.6 to 23.3] | 32.5 [28.7 to 36.8] | 18.4 [16.0 to 21.1] | 35.4 [31.3 to 40.1] | 8.7 [7.5 to 10.0]
  Victoria, POST: number analyzed (Participants) | 425 | 453 | 424 | 447 | 423 | 454 | 259
  Victoria, POST | 194.4 [171.3 to 220.7] | 317.8 [287.1 to 351.8] | 197.4 [175.9 to 221.6] | 301.7 [272.2 to 334.3] | 52.6 [45.2 to 61.2] | 86.6 [77.4 to 96.9] | 127.3 [109.4 to 148.1]
  Yamagata, Day 0: number analyzed (Participants) | 423 | 453 | 423 | 447 | 424 | 453 | 259
  Yamagata, Day 0 | 27.4 [23.8 to 31.7] | 116.2 [102.2 to 132.1] | 29.5 [25.6 to 34.0] | 111.6 [98.3 to 126.8] | 29.5 [25.5 to 34.1] | 139.6 [124.6 to 156.4] | 7.7 [7.0 to 8.6]
  Yamagata, POST | 363.4 [327.8 to 402.9] | 707.5 [648.7 to 771.5] | 103.2 [91.7 to 116.1] | 363.7 [330.4 to 400.3] | 416.7 [374.5 to 463.7] | 787.1 [731.3 to 847.2] | 192.7 [172.1 to 215.7]

7. Secondary Outcome: Number of Subjects Seroconverted Against 4 Strains of Influenza Disease - By Age Strata
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥1:40, or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The vaccine strains assessed were A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Florida/4/2006 (Yamagata) flu strains. Subjects were assessed according to 3 age categories, 3-8 years, 9-17 years and 6-35 months.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 (3-8 Years) Group | GSK2282512A 1 (9-17 Years) Group | Victoria Strain Fluarix (3-8 Years) Group | Victoria Strain Fluarix (9-17 Years) Group | Yamagata Strain Fluarix (3-8 Years) Group | Yamagata Strain Fluarix (9-17 Years) Group | GSK2282512A 2 Group
Number analyzed (Participants) | 423 | 453 | 423 | 447 | 424 | 453 | 259
Participants
  H1N1, POST | 374 | 365 | 390 | 365 | 380 | 370 | 220
  H3N2, POST: number analyzed (Participants) | 423 | 453 | 423 | 447 | 423 | 453 | 259
  H3N2, POST | 291 | 323 | 282 | 308 | 296 | 314 | 189
  Victoria, POST: number analyzed (Participants) | 423 | 453 | 423 | 447 | 423 | 453 | 259
  Victoria, POST | 329 | 324 | 326 | 296 | 133 | 129 | 219
  Yamagata, POST | 366 | 293 | 181 | 178 | 372 | 272 | 243

8. Secondary Outcome: Number of Subjects Seroprotected Against 4 Strains of Influenza Disease - By Age Strata
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition titer ≥ 1:40. The 4 assessed influenza strains were the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Florida/4/2006 flu strains. Subjects were assessed according to 3 age categories, 3-8 years, 9-17 years and 6-35 months.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 (3-8 Years) Group | GSK2282512A 1 (9-17 Years) Group | Victoria Strain Fluarix (3-8 Years) Group | Victoria Strain Fluarix (9-17 Years) Group | Yamagata Strain Fluarix (3-8 Years) Group | Yamagata Strain Fluarix (9-17 Years) Group | GSK2282512A 2 Group
Number analyzed (Participants) | 425 | 453 | 424 | 447 | 424 | 454 | 259
Participants
  H1N1, Day 0: number analyzed (Participants) | 423 | 453 | 423 | 447 | 424 | 453 | 259
  H1N1, Day 0 | 209 | 271 | 218 | 278 | 207 | 270 | 87
  H1N1, POST | 405 | 445 | 412 | 436 | 405 | 443 | 232
  H3N2, Day 0: number analyzed (Participants) | 423 | 453 | 423 | 447 | 423 | 453 | 259
  H3N2, Day 0 | 161 | 134 | 174 | 127 | 168 | 156 | 7
  H3N2, POST | 379 | 437 | 390 | 418 | 389 | 430 | 193
  Victoria, Day 0: number analyzed (Participants) | 423 | 453 | 423 | 447 | 424 | 453 | 259
  Victoria, Day 0 | 144 | 244 | 163 | 241 | 150 | 250 | 28
  Victoria, POST: number analyzed (Participants) | 425 | 453 | 424 | 447 | 423 | 454 | 259
  Victoria, POST | 398 | 440 | 406 | 433 | 271 | 372 | 228
  Yamagata, Day 0: number analyzed (Participants) | 423 | 453 | 423 | 447 | 424 | 453 | 259
  Yamagata, Day 0 | 205 | 373 | 209 | 374 | 220 | 402 | 22
  Yamagata, POST | 419 | 450 | 361 | 444 | 420 | 453 | 250

9. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition Antibodies Against 4 Strains of Influenza Disease - By Age Strata
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0 (i.e. the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer). The 4 assessed influenza strains were the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Florida/4/2006 (Yamagata) flu strains. Subjects were assessed according to 3 age categories, 3-8 years, 9-17 years and 6-35 months.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | GSK2282512A 1 (3-8 Years) Group | GSK2282512A 1 (9-17 Years) Group | Victoria Strain Fluarix (3-8 Years) Group | Victoria Strain Fluarix (9-17 Years) Group | Yamagata Strain Fluarix (3-8 Years) Group | Yamagata Strain Fluarix (9-17 Years) Group | GSK2282512A 2 Group
Number analyzed (Participants) | 423 | 453 | 423 | 447 | 424 | 453 | 259
fold change
  H1N1, POST | 12.50 [11.31 to 13.82] | 12.12 [10.67 to 13.77] | 14.20 [12.83 to 15.71] | 12.52 [11.07 to 14.17] | 14.56 [13.20 to 16.05] | 14.29 [12.52 to 16.31] | 11.95 [10.52 to 13.59]
  H3N2, POST: number analyzed (Participants) | 423 | 453 | 423 | 447 | 423 | 453 | 259
  H3N2, POST | 7.02 [6.30 to 7.84] | 8.91 [7.85 to 10.11] | 6.82 [6.09 to 7.64] | 7.94 [7.02 to 8.97] | 7.29 [6.51 to 8.16] | 8.27 [7.32 to 9.34] | 10.94 [9.64 to 12.42]
  Victoria, POST: number analyzed (Participants) | 423 | 453 | 423 | 447 | 423 | 453 | 259
  Victoria, POST | 10.64 [9.41 to 12.02] | 9.65 [8.42 to 11.07] | 9.75 [8.61 to 11.04] | 9.28 [8.04 to 10.71] | 2.85 [2.58 to 3.16] | 2.44 [2.25 to 2.65] | 14.61 [12.84 to 16.63]
  Yamagata, POST | 13.23 [11.74 to 14.90] | 6.09 [5.42 to 6.84] | 3.49 [3.18 to 3.84] | 3.26 [2.93 to 3.62] | 14.11 [12.57 to 15.84] | 5.63 [5.02 to 6.33] | 24.92 [21.98 to 28.26]

10. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms After Vaccination
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity grade. Grade 3 pain for subjects < 5 years of age = Cried when limb was moved/spontaneously painful; Grade 3 pain for subjects ≥ 5 years of age = Significant pain at rest, pain that preventeded normal everyday activities. Grade 3 redness and swelling were defined as redness/swelling above 100 millimeters (mm).
Time Frame: During the 7-day follow-up period (Days 0-6) after vaccination
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with vaccine administration documented, solely on subjects with symptom sheet completed for the reported specific symptom.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 913 | 912 | 916 | 294
Participants
  Any pain | 637 | 538 | 542 | 148
  Grade 3 pain | 35 | 21 | 26 | 6
  Any redness | 57 | 38 | 36 | 24
  Grade 3 redness | 1 | 0 | 0 | 2
  Any swelling | 64 | 40 | 39 | 18
  Grade 3 swelling | 1 | 0 | 0 | 1

11. Secondary Outcome: Number of Days With Solicited Local Symptoms After Vaccination
Description: Duration was assessed via tabulation of the number of days with local symptoms of any grade after vaccination with Dose 1 and Dose 2 respectively. Solicited local symptoms assessed for duration were pain, redness and swelling.
Time Frame: During the 7-day follow-up period (Days 0-6) after vaccination
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed only on subjects that reported the specific symptom.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 597 | 497 | 510 | 131
Days
  Pain, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Pain, Dose 2: number analyzed (Participants) | 169 | 151 | 141 | 76
  Pain, Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Redness, Dose 1: number analyzed (Participants) | 48 | 29 | 32 | 13
  Redness, Dose 1 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 5.0]
  Redness, Dose 2: number analyzed (Participants) | 13 | 11 | 10 | 14
  Redness, Dose 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0] | 1.5 [1.0 to 3.0] | 2.5 [1.0 to 4.0]
  Swelling, Dose 1: number analyzed (Participants) | 57 | 30 | 35 | 10
  Swelling, Dose 1 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 1.5 [1.0 to 3.0]
  Swelling, Dose 2: number analyzed (Participants) | 12 | 15 | 7 | 11
  Swelling, Dose 2 | 2.5 [2.0 to 4.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 3.0 [2.0 to 4.0]

12. Secondary Outcome: Number of Subjects Below 5 Years of Age With Any, Grade 3 and Related Solicited General Symptoms
Description: Symptoms assessed were drowsiness, irritability, loss of appetite and temperature. Any = Incidence of a particular symptom regardless of intensity grade or relationship to vaccination. Any temperature = Axillary temperature ≥ 38.0 degrees Celsius (°C). Grade 3 temperature = Axillary temperature ≥ 39.0°C. Grade 3 irritability = Crying that could not be comforted/ preventing normal activity. Grade 3 drowsiness = Drowsiness preventing normal activity. Grade 3 loss of appetite = Not eating at all. Related = A general symptom assessed by the investigator as causally related to vaccination.
Time Frame: During the 7-day follow-up period (Days 0-6) after vaccination
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 185 | 187 | 189 | 292
Participants
  Any drowsiness | 46 | 47 | 51 | 102
  Grade 3 drowsiness | 0 | 3 | 1 | 7
  Related drowsiness | 34 | 40 | 42 | 93
  Any irritability | 59 | 44 | 48 | 141
  Grade 3 irritability | 3 | 0 | 3 | 14
  Related irritability | 45 | 36 | 45 | 130
  Any loss of appetite | 40 | 41 | 35 | 93
  Grade 3 loss of appetite | 0 | 6 | 3 | 5
  Related loss of appetite | 21 | 28 | 24 | 73
  Any temperature | 15 | 16 | 15 | 27
  Grade 3 temperature | 3 | 5 | 5 | 6
  Related temperature | 6 | 10 | 6 | 18

13. Secondary Outcome: Number of Subjects 5 Years of Age and Above With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms, headache, joint pain at other location, muscle aches, shivering and temperature. Any = Incidence of a particular symptom regardless of intensity grade or relationship to vaccination. Any temperature = axillary temperature ≥ 38.0 °C. Grade 3 temperature = axillary temperature ≥ 39.0°C. Grade 3 symptom = Symptom that prevented normal activity. Related = A general symptom assessed by the investigator as causally related to vaccination.
Time Frame: During the 7-day follow-up period (Days 0-6) after vaccination
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group
Number analyzed (Participants) | 727 | 725 | 726
Participants
  Any fatigue | 173 | 177 | 177
  Grade 3 fatigue | 6 | 13 | 8
  Related fatigue | 143 | 149 | 134
  Any gastrointestinal symptoms | 80 | 82 | 72
  Grade 3 gastrointestinal symptoms | 9 | 8 | 6
  Related gastrointestinal symptoms | 55 | 51 | 37
  Any headache | 170 | 171 | 157
  Grade 3 headache | 8 | 9 | 10
  Related headache | 134 | 134 | 116
  Any joint pain at other location | 103 | 95 | 81
  Grade 3 joint pain at other location | 4 | 5 | 1
  Related joint pain at other location | 82 | 80 | 67
  Any muscle aches | 222 | 194 | 193
  Grade 3 muscle aches | 6 | 5 | 9
  Related muscle aches | 202 | 178 | 170
  Any shivering | 55 | 51 | 53
  Grade 3 shivering | 4 | 10 | 4
  Related shivering | 45 | 35 | 41
  Any temperature | 26 | 33 | 20
  Grade 3 temperature | 5 | 8 | 2
  Related temperature | 16 | 18 | 13

14. Secondary Outcome: Number of Days With Solicited General Symptoms After Vaccination in Subjects Below 5 Years of Age
Description: Duration was assessed via tabulation of the number of days with local symptoms of any grade after vaccination with Dose 1 and Dose 2, respectively. Solicited general symptoms assessed for duration in subjects below 5 years of age were drowsiness, irritability and loss of appetite.
Time Frame: During the 7-day follow-up period (Days 0-6) after vaccination
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 48 | 37 | 44 | 120
Days
  Drowsiness, Dose 1: number analyzed (Participants) | 39 | 37 | 44 | 85
  Drowsiness, Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Drowsiness, Dose 2: number analyzed (Participants) | 16 | 18 | 17 | 45
  Drowsiness, Dose 2 | 1.0 [1.0 to 1.5] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Irritability, Dose 1: number analyzed (Participants) | 48 | 31 | 41 | 120
  Irritability, Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Irritability, Dose 2: number analyzed (Participants) | 25 | 22 | 16 | 74
  Irritability, Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.5] | 2.0 [1.0 to 3.0]
  Loss of appetite, Dose 1: number analyzed (Participants) | 32 | 30 | 25 | 64
  Loss of appetite, Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Loss of appetite, Dose 2: number analyzed (Participants) | 13 | 15 | 14 | 48
  Loss of appetite, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0] | 3.0 [1.0 to 5.0] | 2.0 [1.0 to 3.0]

15. Secondary Outcome: Number of Days With Solicited General Symptoms After Vaccination in Subjects 5 Years of Age and Above
Description: Duration was assessed via tabulation of the number of days with local symptoms of any grade after vaccination with Dose 1 and Dose 2, respectively. Solicited general symptoms assessed for duration in subjects 5 years of age and above were fatigue, gastrointestinal symptoms, headache, joint pain at other location, muscle aches and shivering.
Time Frame: During the 7-day follow-up period (Days 0-6) after vaccination
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group
Number analyzed (Participants) | 207 | 180 | 179
Days
  Fatigue, Dose 1: number analyzed (Participants) | 161 | 171 | 167
  Fatigue, Dose 1 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Fatigue, Dose 2: number analyzed (Participants) | 27 | 19 | 19
  Fatigue, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Gastrointestinal symptoms, Dose 1: number analyzed (Participants) | 70 | 70 | 65
  Gastrointestinal symptoms, Dose 1 | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 17 | 16 | 9
  Gastrointestinal symptoms, Dose 2 | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Headache, Dose 1: number analyzed (Participants) | 160 | 160 | 146
  Headache, Dose 1 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Headache, Dose 2: number analyzed (Participants) | 20 | 19 | 17
  Headache, Dose 2 | 1.5 [1.0 to 2.5] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Joint pain at other location, Dose 1: number analyzed (Participants) | 94 | 86 | 76
  Joint pain at other location, Dose 1 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 1.5 [1.0 to 3.0]
  Joint pain at other location, Dose 2: number analyzed (Participants) | 21 | 13 | 10
  Joint pain at other location, Dose 2 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Muscle aches, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Muscle aches, Dose 2: number analyzed (Participants) | 44 | 27 | 30
  Muscle aches, Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Shivering, Dose 1: number analyzed (Participants) | 51 | 50 | 50
  Shivering, Dose 1 | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Shivering, Dose 2: number analyzed (Participants) | 8 | 1 | 4
  Shivering, Dose 2 | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 2.0]

16. Secondary Outcome: Number of Days With Fever in All Subjects Regardless of Their Age After Vaccination
Description: Duration for fever was assessed via tabulation of the number of days with local symptoms of fever (axillary temperature ≥ 38°C) after vaccination with Dose 1 and Dose 2, respectively.
Time Frame: During the 7-day follow-up period (Days 0-6) after vaccination
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 25 | 43 | 26 | 16
Days
  Fever, Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Fever, Dose 2: number analyzed (Participants) | 17 | 7 | 9 | 12
  Fever, Dose 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.5]

17. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any unsolicited AE(s) = Occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 unsolicited AE = Occurrence of any unsolicited AE that prevented normal activities. Related unsolicited AE(s) = Occurrence of an unsolicited AE assessed by the investigator to be causally related to vaccination.
Time Frame: During the 28-day follow-up period (Day 0-27) after vaccination
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 932 | 929 | 932 | 301
Participants
  Any unsolicited AE(s) | 283 | 291 | 275 | 160
  Grade 3 unsolicited AE(s) | 40 | 41 | 35 | 24
  Related unsolicited AE(s) | 44 | 47 | 44 | 43

18. Secondary Outcome: Number of Subjects With Any and Related Potential Immune-mediated Diseases (pIMDs) After Vaccination
Description: Potential immune-mediated diseases (pIMDs) are a subset of adverse events that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology.
  Any pIMD(s) = Occurrence of any pIMD(s) regardless of intensity grade or relation to vaccination. Related pIMD(s) = pIMD assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (from Day 0 to Day 180)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 932 | 929 | 932 | 301
Participants
  Any pIMD(s) | 0 | 1 | 1 | 0
  Related pIMD(s) | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Subjects With Any and Related Medically-attended Adverse Events (MAEs) After Vaccination
Description: Medically-attended adverse events (MAEs) were non-serious and serious events leading to an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits. If a medically-attended adverse event was leading to hospitalization (or met any other criterion for serious adverse event (SAE)), it was reported as SAE. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.Relationship to vaccination was not assessed for MAEs.
Time Frame: During the entire study period (from Day 0 to Day 180)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 932 | 929 | 932 | 301
Participants | 346 | 335 | 350 | 147

20. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any SAE(s) = Occurrence of any SAE(s) regardless of intensity grade or relation to vaccination. Related SAE(s)= Occurrence of any SAE(s) assessed by the investigator as causally related to vaccination.
Time Frame: During the entire study period (from Day 0 to Day 180)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Number analyzed (Participants) | 932 | 929 | 932 | 301
Participants
  Any SAE(s) | 3 | 6 | 5 | 7
  Related SAE(s) | 0 | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed from Day 0 to Day 180. Systematically and non-systematically assessed frequent adverse events (AEs) were assessed during a 7-day and 28-day post-vaccination period, respectively.
Description: For the systematically-assessed other non-serious AEs, the number of participants at risk included those from Total Vaccinated cohort whose symptom sheet had been completed.
Arm/Group | GSK2282512A 1 Group | Victoria Strain Fluarix Group | Yamagata Strain Fluarix Group | GSK2282512A 2 Group
Serious Adverse Events (participants affected / at risk) | 3/932 | 6/929 | 5/932 | 7/301
Other Adverse Events (participants affected / at risk) | 731/932 | 666/929 | 659/932 | 233/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2282512A 1 Group (N=932) | Victoria Strain Fluarix Group (N=929) | Yamagata Strain Fluarix Group (N=932) | GSK2282512A 2 Group (N=301)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK2282512A 1 Group (N=932) | Victoria Strain Fluarix Group (N=929) | Yamagata Strain Fluarix Group (N=932) | GSK2282512A 2 Group (N=301)
Pain (General disorders) | 637/913 | 538/912 | 542/916 | 148/294
Redness (General disorders) | 57/913 | 38/912 | 36/916 | 24/294
Swelling (General disorders) | 64/913 | 40/912 | 39/916 | 18/294
Drowsiness (General disorders) | 46/185 | 47/187 | 51/189 | 102/292 — Assessed in subjects less than 5 years of age in all study Groups.
Irritability (General disorders) | 59/185 | 44/187 | 48/189 | 141/292 — Assessed in subjects less than 5 years of age in all study Groups.
Loss of appetite (General disorders) | 40/185 | 41/187 | 35/189 | 93/292 — Assessed in subjects less than 5 years of age in all study Groups.
Temperature (General disorders) | 15/185 | 16/187 | 15/189 | 27/292 — Assessed in subjects less than 5 years of age in all study Groups.
Fatigue (General disorders) | 173/727 | 177/725 | 177/726 | 0/0 — Assessed in subjects 5 years of age and above in GSK2282512A 1 Group, Victoria strain Fluarix Group and Yamagata strain Fluarix Group.
Gastrointestinal (General disorders) | 80/727 | 82/725 | 72/726 | 0/0 — Assessed in subjects 5 years of age and above in GSK2282512A 1 Group, Victoria strain Fluarix Group and Yamagata strain Fluarix Group.
Headache (General disorders) | 170/727 | 171/725 | 157/726 | 0/0 — Assessed in subjects 5 years of age and above in GSK2282512A 1 Group, Victoria strain Fluarix Group and Yamagata strain Fluarix Group.
Joint pain at other location (General disorders) | 103/727 | 95/725 | 81/726 | 0/0 — Assessed in subjects 5 years of age and above in GSK2282512A 1 Group, Victoria strain Fluarix Group and Yamagata strain Fluarix Group.
Muscle aches (General disorders) | 222/727 | 194/725 | 193/726 | 0/0 — Assessed in subjects 5 years of age and above in GSK2282512A 1 Group, Victoria strain Fluarix Group and Yamagata strain Fluarix Group.
Shivering (General disorders) | 55/727 | 51/725 | 53/726 | 0/0 — Assessed in subjects 5 years of age and above in GSK2282512A 1 Group, Victoria strain Fluarix Group and Yamagata strain Fluarix Group.
Upper respiratory tract infection (Infections and infestations) | 36 | 30 | 33 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 53 | 38 | 49 | 34
Nasopharyngitis (Infections and infestations) | 48 | 47 | 43 | 14
Pyrexia (General disorders) | 19 | 16 | 13 | 21
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 17 | 12 | 19 | 33
Diarrhoea (Gastrointestinal disorders) | 11 | 10 | 7 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.